CLINICAL TRIAL: NCT04989036
Title: Clinical and Radiographic Evaluation of Apexogenesis Using Calcium Hydroxide Pulpotomy Versus Calcium Silicate-Based Material (Biodentine™) Pulpotomy in Cariously Exposed Vital Immature Permanent First Molars: A Randomized Controlled Trial With 12 Months Follow Up
Brief Title: Biodentine Vital Pulpotomy in Immature Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shereen H Elshamy, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 842014
Record Dates: First submitted 2021-06-24; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Pulp Exposure, Dental
MeSH Terms: conditions — Dental Pulp Exposure | interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT), parallel group with 1:1 allocation ratio and equivalence framework. Triple blinded (patient, radiographic assessors of results and statistician) Ethics approval by the Human Research Ethics committee at Faculty of Dentistry- Cairo University was taken.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blinded (patient, radiographic assessors of results and statistician)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALCIUM HYDROXIDE™ (Experimental): Non-setting Calcium hydroxide Pulpotomy capping agent. Deepak. Promotion Industrial Park, Bari Brahmana, Jammu - 181133 India form : powder and liquid. application : Calcium hydroxide was mixed with saline to a thick consistency immediately before use. The paste was carefully placed on the pulp stump surface 2-3 mm thick over a small sterile wet cotton with a small condenser, and the excess material was scraped off.
  Interventions: Procedure: pulpotomy
- Biodentine ™ (Experimental): Biodentine ™ Pulpotomy capping agent. Calcium Silicate-Based Material.Septodent®, Saint-Maurdes-Fosses, France form: capsule and liquid. application: According to the instructions of manufacture, Biodentine ™powder and liquid were mixed to achieve a creamy consistency, by mixing a single-unit powder part and 5 drops of a single-unit liquid part for 30 seconds by mixing device . Final mixing and adjustment were done manually to obtain the desired consistency for each case
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: pulpotomy — Pulpotomy refers to the removal of the entire coronal pulp to the level of the root canal orifice(s) or as much as 2-3 mm apical to the orifices. Pulpotomy has indications similar to those of a partial pulpotomy except that the pulp in question is likely to have more extensive inflammation. Since pulpal inflammation is unlikely to extend past the canal orifices, pulpotomy is similar to a partial pulpotomy except that the entire mass of coronal pulp tissue is removed
  Other Names: vital pulp therapy; apexogensis

SUMMARY:
This study aimed to evaluate the clinical and radiographic success of pulpotomy in cariously exposed vital immature first permanent molars using calcium hydroxide and calcium silicate-based material (Biodentine ™). After a 12 months postoperative period, Biodentine ™ proved very useful as a successful pulpotomy agent in young permanent teeth.

DETAILED DESCRIPTION:
Objective: This study aimed to evaluate the clinical and radiographic success of pulpotomy in cariously exposed vital immature first permanent molars using calcium hydroxide and calcium silicate-based material (Biodentine ™).

Participants and methods:

This study was carried out on patients attending an outpatient clinic in Pediatric Dentistry and Dental Public Health Department - Faculty of Dentistry - Cairo University - Egypt. A total of thirty-five patients had thirty-eight vital immature first permanent molar with deep caries, who satisfied the eligibility criteria and completed the follow-up period. Their age ranged between six years to nine years old with a mean age of 7.5+/-1 years. All teeth were mandibular. In this study, pulpotomy was performed to preserve the vitality and function of the remaining radicular pulp tissue, followed by applying one of the investigated pulp capping materials.

ELIGIBILITY:
Inclusion Criteria:

* Medical history: Healthy children with no physical or mental disorders assured through medical history questioning.
* Mandibular vital immature first permanent molar with deep caries. Restorable. No clinical evidence of extensive pulp degeneration or periapical pathology.No radiographic evidence of periapical pathosis or interradicular bone loss, internal/external resorption and pulp calcification.

Exclusion Criteria:

* 1. Patients refuse to cooperate. 2. Spontaneous pain or severe pain which doesn't stop with analgesics. 3. Hemorrhage control wasn't achievable at the operative procedures

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pain severity | 12 months
  ordinal outcome measured with direct questioning to the patient using Verbal Rating Scale ( VRS)
Absences of swelling / fistulous tract | 12 months
  binary outcome observed clinically

SECONDARY OUTCOMES:
Absence of tenderness to percussion | 12 months
  binary outcome detected by back of mirror
Absence of internal or external root resorption | 12 months
  binary outcome detected in periapical radiograph
Root maturation | 12 months
  binary outcome detected in periapical radiograph

IPD SHARING:
Plan to Share IPD: Yes
after publication , sharing all the data with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 year
Access Criteria: after publication